CLINICAL TRIAL: NCT02362490
Title: HBsAg Clearance of Peginterferon Treatment in Patients Who Had Chronic Hepatitis B and Were on the Treatment of Nucleoside(Acid) Analogues
Brief Title: Efficacy of Peginterferon Alpha 2a Therapy in Chronic Hepatitis B Patients Being Treated With Nucleoside(Acid) Analogues
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTXY004
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; interferon; Nucleotide analogues; HBsAg
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- peginterferon alpha 2a (Experimental): in this group, patients who were on treatment of Nucleoside (Acid) Analogues and had achieved HBsAg level ≤250 IU/ml will switch to treatment of peginterferon alpha 2a for 72 week.
  Interventions: Drug: peginterferon alpha 2a
- control group (No Intervention): in this group, patients who were on treatment of Nucleoside(Acid) Analogues and had achieved HBsAg level ≤250 IU/ml will be continue to treatment of Nucleoside(Acid) Analogues for 72 week.

INTERVENTIONS:
Drug: peginterferon alpha 2a — in this group,patients will receive 180 ug of peginterferon alpha 2a injection weekly for 72 weeks
  Other Names: PEG-IFN a-2a
  Arms: peginterferon alpha 2a

SUMMARY:
Antiviral therapy is the most important method to slow and stop the progress of the disease in patients with chronic hepatitis B (CHB). Nucleoside (acid) analogues (NA) can Effectively suppress HBV replication, but it should be continue used and relapse would happen in most patients after withdrawal of therapy. However, long-term use of NA could induce viral resistance mutation lead to loss of efficacy. Interferon treatment can enhance specific and non-specific immune function in chronic hepatitis B patients, make patients get immune control to HBV infection and obtain sustained response after treatment. Thus the CHB patients on the treatment of NA should be stop NA treatment after interferon treatment. In this study, the effects of interferon treatment in CHB patients who were on the NA treatment and obtained HBsAg level≤250 IU/ml.

DETAILED DESCRIPTION:
In this trial, patients who were CHB and treated with NA more than 6 months, still on the treatment and achieved HBsAg level ≤250 IU/ml with HBV DNA undetectable will be randomized enrolled into group A (Intervention group), in which patients switch to interferon therapy for 72 weeks, group B(control group), patients continue treated with NA for 72 weeks. Serum HBV DNA load, HBsAg/anti-HBs level, HBeAg/anti-HBe will be tested at enrollment and every 3 months during the treatment course. Parameters of Liver and kidney function, and liver ultrasound examination will be tested with intervals 1-3 months. The efficacies of interferon treatment were devalued by the rate of HBsAg clearance and decline of HBsAg levels on the 72 weeks of interferon treatment compared with control group.

ELIGIBILITY:
Inclusion Criteria:

* patients who were chronic hepatitis B and had achieved HBsAg level ≤250 IU/ml on treatment of Nucleoside (acid) Analogues

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
rate of HBsAg loss | 72 weeks
  the effects of peginterferon alpha 2a will be evaluated by HBsAg loss defined as HBsAg level lower than 0.05 IU/ml after 72 week treatment,compared control group.

SECONDARY OUTCOMES:
decline of HBsAg level | 72 weeks
  secondary outcome was evaluated by the decline of HBsAg level after 72 weeks of peginterferon alpha 2a treatment compared with control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan hospital,Capital Medical University, Beijing, Beijing Municipality, China